CLINICAL TRIAL: NCT02101073
Title: A Phase I, Open-Label Study Evaluating the Bioavailability of ALX-0061 After Subcutaneous and Intravenous Administration in Healthy Volunteers.
Brief Title: ALX-0061 Phase I Bioavailability Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ablynx, a Sanofi company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALX0061-C102; 2013-005493-21 (EudraCT Number)
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ALX-0061

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- ALX-0061 low dose i.v. (Experimental)
  Interventions: Biological: ALX-0061
- ALX-0061 high dose i.v. (Experimental)
  Interventions: Biological: ALX-0061
- ALX-0061 low dose s.c. (Experimental)
  Interventions: Biological: ALX-0061
- ALX-0061 middle dose s.c. (Experimental)
  Interventions: Biological: ALX-0061
- ALX-0061 high dose s.c. (Experimental)
  Interventions: Biological: ALX-0061

INTERVENTIONS:
Biological: ALX-0061 — single dose, intravenous
  Arms: ALX-0061 high dose i.v.; ALX-0061 low dose i.v.
Biological: ALX-0061 — single dose, subcutaneous
  Arms: ALX-0061 high dose s.c.; ALX-0061 low dose s.c.; ALX-0061 middle dose s.c.

SUMMARY:
The overall aims of the study are:

* To assess the bioavailability of single doses of ALX-0061, administered s.c. at three dose levels, using 2 corresponding single i.v. dose levels as reference.
* To provide additional information on pharmacokinetics and pharmacodynamics of ALX-0061.
* To further determine the safety and tolerability of ALX-0061.
* To further evaluate the systemic (serum) immunogenicity of ALX-0061.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy volunteers.
2. Gender: male or female.
3. Age 18 to 55 years.
4. Body mass index (BMI): 18.0 ≥ BMI < 30.0 kg/m2.

Key Exclusion Criteria:

1. Any active inflammatory condition, or autoimmune disorder such as lupus erythematosus, multiple sclerosis or rheumatoid arthritis (RA).
2. Any current or recent (within 4 weeks prior to dose) signs or symptoms of infection that requires parenteral antibiotic administration.
3. Symptomatic infection, or suspicion thereof in the last 1 week prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2014-07-31 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: serum concentration of ALX-0061 after single subcutaneous (s.c.) and single intravenous (i.v.) doses of ALX-0061 in healthy volunteers | Day 1 to Day 32 +/- 2 days after dosing for low dose treatment arms, Day 1 to Day 46 +/-2 days after dosing for middle dose treatment arm, Day 1 to Day 53 +/- 2 days after dosing for high dose treatment arms

SECONDARY OUTCOMES:
Pharmacodynamics: concentration in plasma of total soluble Interleukin-6 receptor (sIL-6R) and in serum of IL-6 | During screening untill final visit (i.e. 60 +/- 2 days after dosing for the low dose and middle dose treatment arms and 83 +/- 2 days after dosing for the high dose treatment arms)
Safety and tolerability: safety markers | From signing of informed consent until final visit (i.e. 60 +/- 2 days for the low dose and middle dose treatment arms and 83 +/- 2 days for the high dose treatment arms
  * Adverse events and concomitant medication
  * Clinical laboratory
  * Vital signs
  * 12-lead ECG
  * Physical examination
  * Local reactions
Immunogenicity: concentration of Anti-Drug Antibodies (ADA) in serum | From screening until final visit (i.e. 60+/- 2 days after dosing for the low dose and middle dose treatment arms and 83 +/- 2 days after dosing for the high dose treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Steven De Bruyn, MD, Study Director — Ablynx NV
Locations (1):
- Zuidlaren, Netherlands